CLINICAL TRIAL: NCT03000218
Title: Clinical Study Evaluating Pharmacokinetics and Biomarkers After Ursodeoxycholic Acid (UDCA) Administration to Subjects Who Are Overweight and Have Liver Problems
Brief Title: Evaluation of PK and Biomarkers After UDCA Administrations to Subjects Who Are Overweight and Have Liver Problems
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae Yong Chung, MD, PhD, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDCA_overweight_LFTabnormal
Record Dates: First submitted 2016-06-21; First posted 2016-12-21 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Overweight; Abnormal Liver Function Tests
MeSH Terms: conditions — Overweight | interventions — Ursodeoxycholic Acid; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- UDCA 8 wks (Experimental): Day 1 to 56: Ursodeoxycholic acid 300mg bid
  Interventions: Drug: Ursodeoxycholic acid
- UDCA for 4wks/UDCA+metformin for 4wks (Experimental): Day 1 to 28: Ursodeoxycholic acid 300mg bid Day 29 to 56: Ursodeoxycholic acid 300mg and Metformin 500mg bid
  Interventions: Drug: Ursodeoxycholic acid; Drug: Metformin
- Placebo (Placebo Comparator): Day 1 to 56: Placebo bid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ursodeoxycholic acid — Ursodeoxycholic acid 300mg bid for 8 weeks
  Other Names: Ursa tab
  Arms: UDCA 8 wks; UDCA for 4wks/UDCA+metformin for 4wks
Drug: Metformin — Day 29 to 56: Metformin 500mg bid
  Other Names: Diabex tab
  Arms: UDCA for 4wks/UDCA+metformin for 4wks
Drug: Placebo — Day 1 to 56: Placebo bid
  Arms: Placebo

SUMMARY:
A clinical study to evaluate pharmacokinetics, metabolomics and biomarker in subjects who are overweight and have liver problems after ursodeoxycholic acid multiple administration

DETAILED DESCRIPTION:
This study has a randomized, open-label, three-treatment, one-sequence, placebo-controlled, multiple drug administration design. The purpose of this study is as follows; To evaluate pharmacokinetics, metabolomics and biomarker in subjects who are overweight and have liver problems after ursodeoxycholic acid administration

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects aged 18 - 50 years
* A body mass index (BMI) in the range of 25.0 kg/m2 - 30.0 kg/m2.
* A alanine aminotransferase (ALT) in the range of 40 - 200 IU/L
* Good health based on complete medical history, physical examinations, vital signs, electrocardiography (ECG), and clinical laboratory evaluations.

Exclusion Criteria:

* Subjects who have clinically significant disease of cardiovascular, respiratory, renal, endocrinological, hematological, gastrointestinal, neurological(central nervous system), psychiatric disorders or malignant tumor
* Subject judged not eligible for study participation by investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of ursodeoxycholic acid | Day 1, 15, 29, 57 predose (0h), Day 29 1, 2, 3, 4h
Change from Baseline Low-density lipoprotein cholesterol at 8 weeks | Day 1, 29, 57, 71 predose (0h)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Yong Chung, M.D., Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided